CLINICAL TRIAL: NCT06452290
Title: PET Biomarker Study for Antidepressant Response Prediction in Major Depressive Disorder
Acronym: TEPDEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Antoine VERGER, Principal Investigator, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024PI076
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brain 18F-FDG PET-CT (Experimental): The strategy under investigation is a medical device: a PET/CT scanner using the radiopharmaceutical 18F-FDG.
  Interventions: Device: brain 18F-FDG PET-CT

INTERVENTIONS:
Device: brain 18F-FDG PET-CT — PET scanner, Philips VEREOS PET/CT scanner. Three Philips VEREOS digital PET/CT scanners are installed in the nuclear medicine department.

SUMMARY:
Major depressive disorder has a prevalence of 4.7% in the general population and is ranked as the leading cause of disability worldwide. The efficacy of current antidepressants is limited, as 50-60% of patients do not achieve a sufficient response to treatment : 12% achieve only a partial response, while 19-34% do not respond at all. These uncertain clinical effects are only observed after several weeks of treatment. For better patient management, there is an urgent need to identify markers for predicting and monitoring therapeutic response.

Psychiatrists at the Nancy Psychotherapeutic Center are about to launch a "MESANTIDEP" study, in which they will evaluate the electroretinogram (ERG) as a biomarker for predicting and monitoring therapeutic response.

The TEPDEP study described in this protocol would evaluate 18F-FDG brain PET/CT as a biomarker for predicting antidepressant response in a treatment-naive patient population.

It is planned to offer the PET/CT study to patients included in the SSRI arm of the MesantiDEP study.

The hypothesis of this study is that 18F-FDG PET/CT could be a biomarker for predicting response to selective serotonin reuptake inhibitor (SSRI) antidepressants.

DETAILED DESCRIPTION:
Major depressive disorder has a prevalence of 4.7% in the general population and is ranked as the leading cause of disability worldwide . The efficacy of current antidepressants is limited, as 50-60% of patients do not achieve a sufficient response to treatment: 12% achieve only a partial response, while 19-34% do not respond at all . These uncertain clinical effects are only observed after several weeks of treatment . For better patient management, there is an urgent need to identify markers for predicting and monitoring therapeutic response.

Psychiatrists at the Nancy Psychotherapeutic Center are about to launch a "MESANTIDEP" study, in which they will evaluate the electroretinogram as a biomarker for predicting and monitoring therapeutic response.

In the literature, numerous studies have shown a pattern of carbohydrate hypometabolism characteristic of depression, identified by 18F-FDG brain PET/CT scans. Cerebral metabolism patterns predictive of antidepressant response have also been demonstrated in some clinical trials, with hypermetabolism of the anterior cingulate in responders; and more severe hypometabolism of the anterior cingulate , dorsolateral prefrontal cortex and premotor area in non-responders. However, the studies in the literature group together very heterogeneous populations, with a large proportion of patients not naïve to antidepressant treatment.

The TEPDEP study described in this protocol would evaluate Positons Eission Tomography (PET) with flurodeoxyglucose labelled with fluor-18 (18F-FDG) brain as a biomarker for predicting antidepressant response in a treatment-naive patient population.

It is planned to offer the PET/CT study to patients included in the SSRI arm of the MesantiDEP study.

The hypothesis of this study is that 18F-FDG PET/CT could be a biomarker for predicting response to selective serotonin reuptake inhibitor (SSRI) antidepressants.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 and over, included in the MESANTIDEP study for whom SSRI ( Selective serotonin reuptake inhibitor) treatment is planned.
* Patient who has received full information on the organization of the research and has given written informed consent (or a third person, independent of the investigator and sponsor, in the event of inability to read or write),
* Patient affiliated to a social security scheme or beneficiary of such a scheme

Exclusion Criteria:

* Contraindications for 18F-FDG PET/CT scans
* Presence of chronic neurological or psychiatric pathologies pre-Covid-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Quantitative voxel-by-voxel analysis | 24 months
  Quantitative voxel-by-voxel analysis of cerebral glycolytic metabolism on a group scale

SECONDARY OUTCOMES:
assessing the patient's acceptability of the imaging examination | 24 months
  satisfaction survey
Volumes and topographies of brain regions | 24 months
  Volumes and topographies of brain regions , defined as those showing decreased glycolytic metabolism in 18F-FDG brain PET/CT in relation to quantitative electroretinogram parameters.
Number of possible reclassification | 24 months
  Number of possible reclassification of response to Selective Serotonin Reuptake Inhibitors, by adding 18F-FDG brain PET/CT to electroretinogram